CLINICAL TRIAL: NCT04510376
Title: A Safety Study to Assess the Allergy Potential of Omeza Collagen Matrix in Human Subjects Using the Skin Prick Method
Brief Title: Allergy Potential of Omeza Collagen Matrix in Human Subjects Using the Skin Prick Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omeza, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OMZPRI1F
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Allergic Reaction
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Test article (Experimental)
  Interventions: Device: Test Article
- Histamine Positive Skin Test Control (Active Comparator)
  Interventions: Other: Positive Control
- Aqueous Negative Control (Placebo Comparator)
  Interventions: Other: Negative Control

INTERVENTIONS:
Device: Test Article — Omeza Collagen Matrix
  Arms: Test article
Other: Positive Control — 1.0 mg/mL Histamine Base
  Arms: Histamine Positive Skin Test Control
Other: Negative Control — Aqueous Negative Control
  Arms: Aqueous Negative Control

SUMMARY:
Single-center, monadic, one day study utilizing the skin prick method to assess the allergy potential of Omeza Collagen Matrix in Human Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged 18 years of age and older as demonstrated by selfreported medical history, concurrent medication, and a brief dermal skin assessment of the test sites;
2. Fully informed of the risks of entering the study and willing to provide written informed consent and HIPAA authorization to disclose protected health information;
3. Subject has normal healthy skin on the either volar forearm.

Exclusion Criteria:

Subjects must be excluded if any of the following conditions exist:

1. Self-reported pregnant or nursing at the screening visit;
2. Clinically significant skin disease which may contraindicate participation, including psoriasis, eczema, atopic dermatitis, and active cancer;
3. History of drug abuse or current drug user;
4. Treatment with antihistamine or steroid (any route) administered within the last 7 days;
5. History of anaphylaxis to matrix ingredients (e.g. fish, palm oil, hemp oil, beeswax);
6. Persistent severe/ unstable asthma;
7. Subjects on beta blockers and/or ACE inhibitors;
8. Medical condition which in the opinion of the Investigator would compromise the safety of the subject or confound study results (Subjects with the following conditions: chronic renal failure, CVA, cancer, spinal cord injury, diabetic neuropathy, recent anaphylaxis, limbs affected by lymphoedema, paralysis, or neurogenic abnormalities;
9. Diabetic (type 1 or 2);
10. Subjects taking the following: Antidepressants such as doxepin, other tricyclics, Phenothiazines, and tetracyclics within the last two weeks;
11. Subjects taking OTC cold and flu remedies, "sinus" analgesics, antitussives, antiemetics, sedatives, relaxants, migraine prophylactics (cyproheptadine, pizotifen);
12. Prolonged use of topical corticosteroids;
13. Use of topical moisturizers on the volar forearms;
14. Dermographism "writing on the skin" - common localized hive reaction, characterized by the abrupt onset of welts and hives where the skin is exposed to pressure, scratching, itching, or stroking;
15. Investigator deems the subject an unsuitable candidate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
Allergic Reaction | 20 minutes
  Response of at least 3-mm diameter (with equivalent erythema) more than negative control is required as proof of presence of cutaneous allergen specific IgE

SECONDARY OUTCOMES:
Allergic Reaction | 60 minutes
  Latent reaction to skin prick (safety assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Ellis, M.D., Principal Investigator — PCR Corp; Lori Decaro, Study Director — PCR Corp
Locations (1):
- PCR Corp, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Allergy Diagnostic Testing: An Updated Practice Parameter — https://www.aaaai.org/Aaaai/media/MediaLibrary/PDF%20Documents/Practice%20and%20Parameters/allergydiagnostictesting.pdf